CLINICAL TRIAL: NCT05678829
Title: A Different Method in Reproductive Health and Family Planning: "Virtual Reality Application''
Brief Title: Reproductive Health and Family Planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sümeyye Betül SÖNMEZ (Other Government)
Responsible Party: Sponsor-Investigator, Sümeyye Betül SÖNMEZ, Principal Investigator, Erzurum Regional Training & Research Hospital
Organization: Erzurum Regional Training & Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: betul25
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Virtual Reality; Reproductive Health
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): Using a virtual reality application based on individuals in Virtual Reality creatures, it will be explained for an average of 20 minutes in a time period where they are appropriate, through extensive trainings according to what is given.
  Interventions: Other: Education
- Face to face (Experimental): By using the training room of the family health center specified for the individuals in the Face to face group, training content covering the subjects of reproductive and health and family planning methods will be prepared, and the days when women are suitable will be determined, and each training will be given for 40 minutes with face-to-face classical training method. Educational subjects will be continued in parallel with Virtual Reality group by using Ministry of Health hand brochures and training materials for Face to face group.
  Interventions: Other: Education
- Control (No Intervention): No intervention will be made to the control group during the training.

INTERVENTIONS:
Other: Education — The trainings for the Virtual Reality group will continue in accordance with the training titles according to the weeks, using virtual reality glasses.
  Other Names: virtual reality
  Arms: Face to face; Virtual Reality

SUMMARY:
The aim of this study is to measure the knowledge and attitude levels of women who play a key role in society on reproductive health and family planning, and to determine the changes in their attitudes and behaviors after face-to-face training with virtual reality application.

DETAILED DESCRIPTION:
In a three-month period, using the virtual reality application prepared for the individuals in the Experimental 1 group, it will be explained for an average of 40 minutes in a time period where they are suitable, through the trainings prepared according to the subjects. The literature will be scanned and appropriate educational materials will be created, and animations will be used to support education. The trainings for the Experiment 1 group will continue in accordance with the training titles according to the weeks, using virtual reality glasses. Modern family planning methods will be shown in detail through virtual reality glasses, three dimensions of the methods will be shown and supported by videos.

By using the training room of the family health center specified for the individuals in the Experimental 2 group, training content covering the subjects of reproductive and health and family planning methods will be prepared, and the days when women are suitable will be determined, and each training will be given for 40 minutes with face-to-face classical training method. Educational subjects will be continued in parallel with Experiment 1 group by using Ministry of Health hand brochures and training materials for Experiment 2 group.

ELIGIBILITY:
Inclusion Criteria:

-Being over 20 years old

* Married,
* Being literate,
* Not using modern family planning methods

Exclusion Criteria:

-Being under 20 years old

* not being married
* Not volunteering to participate in the study
* Using modern family planning method
* Not being able to attend the trainings at any stage of the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Married Women's Reproductive Health Protective Attitudes Scale | two week
  Married Women's Reproductive Health Protective Attitudes Scale was developed by Demirci and Karanisoğlu in 2004 to determine the reproductive health protective attitudes and behaviors specific to married women in our country.Married Women's Reproductive Health Protective Attitudes Scale; It is a Likert-type scale, scored between 1 and 5, consisting of 39 easy-to-understand items that women can answer on their own. A minimum of 39 and a maximum of 195 points can be obtained from the scale.Expressing their practices related to their attitudes and behaviors towards protecting their reproductive health according to their frequency and reading each item appropriate for them" "1=Never, 2=Rarely (Very Rarely), 3=Sometimes, 4=Oftentimes and 5=Always" They were asked to select one of the "/regular" options. In this scale, items 5, 10, 16 and 28 were reverse scored.
Family Planning Scale | Two week
  "Family planning attitude scale is a Likert-type scale consisting of 34 items and scored between 1-5. In this easy-to-understand scale, "I totally agree" receives 1 point, "I agree 2 points", "I am undecided 3 points", "I disagree 4 points", "I totally disagree 5 points". There is no item in the scale that needs to be reverse coded.
  A minimum of 34 and a maximum of 170 points can be obtained from the scale. Again, the raw score of each sub-dimension is obtained by summing the items under the sub-dimension. As the total and sub-dimension scores obtained from the scale increase, women's attitudes towards family planning also develop positively.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Betül Sönmez, Study Chair — Ataturk University
Locations (1):
- Ataturk Unıversity, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No